CLINICAL TRIAL: NCT02808481
Title: FOLLOW HEART TRANSPLANT FOR ACHIEVING THE HEART PRIMITIVE RELATED SCLERODERMA SYSTEMIC
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 6410
Record Dates: First submitted 2016-06-17; First posted 2016-06-21 (Estimated); Last update posted 2016-06-21 (Estimated); Status verified 2016-05

CONDITIONS: Systemic Sclerosis
Keywords: systemic sclerosis; cardiac disease; Heart transplantation; primitive cardiac damage
MeSH Terms: conditions — Scleroderma, Systemic; Heart Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Systemic sclerosis is a rare disease. The early cardiac disease affects 10% of patients sclérodemiques.

Heart transplantation in the early cardiac involvement in systemic sclerosis is exceptional.

we see patient data analysis with systemic sclerosis who used cardiac transplantation to understand the primitive cardiac damage associated with systemic sclerosis

ELIGIBILITY:
Inclusion criteria:

* Adult patients meet the criteria for classification of systemic sclerosis
* Adverse primitive heart that required a heart transplant
* Patients who have given their verbal agreement to use their data for research purposes.

Exclusion criteria:

* Localized Scleroderma or sclerodermiform syndrome
* Heart disease secondary to pulmonary or renal impairment
* Refusal to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with systemic sclerosis who used cardiac transplantation for primary cardiac involvemen
Sampling Method: Probability Sample
Enrollment: 9 (Estimated)
Dates: Start 2016-06; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Analysis of data from patients with systemic sclerosis who used cardiac transplantation for primary cardiac involvement | 1month post-transplantation

IPD SHARING:
Plan to Share IPD: No